CLINICAL TRIAL: NCT01951560
Title: A Phase 1, Single Ascending Dose, Double Blind, Placebo Controlled Study to Evaluate the Safety and Tolerability of Valproic Acid in Healthy Volunteers (Part 1) or Trauma Patients(Part 2)
Brief Title: A Study to Evaluate the Safety and Tolerability of Valproic Acid in Healthy Volunteers (Part 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Hasan Alam (Other)
Responsible Party: Sponsor-Investigator, Dr. Hasan Alam, Hasan Alam, MD, Norman Thompson Professor of Surgery Section Head, General Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VPA-C-002
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Shock,Hemorrhagic
MeSH Terms: conditions — Shock, Hemorrhagic | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- valproic acid (Depacon) (Experimental): Valproic acid by IV infusion over one hour
  Interventions: Drug: Valproic Acid
- Isotonic saline solution (Placebo Comparator): The placebo administered by IV infusion over 1 hour
  Interventions: Drug: Isotonic saline solution

INTERVENTIONS:
Drug: Valproic Acid — By infusion over 1 hour
  Other Names: Depacon
  Arms: valproic acid (Depacon)
Drug: Isotonic saline solution — By infusion over 1 hour
  Arms: Isotonic saline solution

SUMMARY:
The purpose of the first part of this study is to determine the safety and tolerability of ascending doses of valproic acid (also known as Depacon) administered as intravenous infusion (IV) in doses ranging from 15 mg/kg to 250 mg/kg in healthy subjects.

The second part of the study will also be to determine the safety and tolerability of single ascending doses of valproic acid administered as IV in trauma subjects with hemorrhagic shock.

DETAILED DESCRIPTION:
Part 1 of the study will be a single center study intended to assess the safety and tolerability of valproic acid dosages at 15 mg/kg, 30 mg/kg, 60 mg/kg, 90 mg/kg, 120 mg/kg, 150 mg/kg 180 mg/kg, 210 mg/kg and 250 mg/kg. Up to 72 healthy subjects (9 dose groups of 8 subjects) will receive single doses of valproic acid or placebo via a 60-min IV infusion in a ratio of 3:1 active drug: placebo.

Part 2 of the study will be a multicenter, double blind, placebo-controlled study in trauma patients with hemorrhagic shock who are able to give consent or severe trauma patients with hemorrhagic shock in whom a legally authorized representative can give consent. Up to 12 patients (2 dose groups of 6 patients) will receive single doses of valproic acid or placebo via a 60-min IV infusion in a ratio of 2:1 active drug : placebo. The dose levels in Part 2 will be the two highest doses that are demonstrated to have acceptable safety profile based on the review of safety data from Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers between the ages of 18 and 65 years, inclusive, in good health based on medical history, physical examination, ECG, and routine laboratory tests (blood chemistry, hematology, urinalysis, and drug screen).
2. Female subjects must be surgically sterilized or postmenopausal. Criteria for menopause are surgical menopause (hysterectomy, oophorectomy) or age > 45 years with absence of menses for greater than 12 months or a serum follicle stimulating hormone (FSH) elevation > 25m IU/mL.(mIU/mL is the unit used to measure human chorionic gonadotropin (hCG) in pregnancy test). Tubal ligation with menses within the past 12 months is not considered to be surgical sterilization.
3. Negative urine pregnancy test in female volunteers
4. Body mass index (BMI) between 18 kg/m2 and 30 kg/m2
5. Subjects must be non-smokers
6. Negative alcohol screen
7. Willing and able to be confined to the clinical research facility as required by the protocol.
8. Willing and able to comply with the investigational nature of the study and able to communicate well with investigators.
9. Ability to comprehend and willingness to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

1. Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies; however, subjects with untreated, asymptomatic, seasonal allergies may be enrolled).
2. Subjects with a-amylase >130 U/L or lipase >300 U/L or creatinine > upper limit of normal (ULN)
3. Subjects with >2times ULN aspartate aminotransferase (AST) or alanine amino transferase (ALT) or >1.5 times total bilirubin
4. Subjects whose screening ECG demonstrates at least one of the following: heart rate > 100 bpm for more than 30 minutes, (the combination of three of the graphical deflections seen on a typical ECG is called the(QRS)) > 120 msec, corrected QT interval (QTc) > 440 msec if male or 450 msec if female, prevalence rate (PR) > 220 msec or any rhythm other than sinus rhythm, sinus bradycardia (HR <40 bpm), or sinus arrhythmia.
5. Subjects with a history of alcohol consumption exceeding 14 drinks/week on average within the 6 months before study entry.
6. Subjects whose sitting blood pressure is above 140/90 mmHg on 2 evaluations at least 10 minutes apart at screening.
7. Subjects who have donated blood in excess of 500 mL within 60 days prior to the first dose of study medication.
8. Subjects with a positive result on drug screen, hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or human immunodeficiency (HIV) tests
9. Subjects who have used prescription or non-prescription drugs, vitamins, herbal supplements or dietary supplements within 14 days prior to the first dose of study medication. Subjects who have used acetaminophen at doses of < 2 grams/day will be eligible for study entry.
10. Subjects who have been treated with an investigational drug within 30 days.
11. Subjects who have previously received or are currently taking valproic acid.
12. Subjects who have a history of drug abuse.
13. Subjects who are not willing to abstain from consuming products containing caffeine (including chocolate), methyl xanthine, or alcohol from Day -1 through the end of the pharmacokinetics (PK) study (day 4 for part 1 subjects).
14. Subjects who have had a febrile illness within 5 days prior to the first dose of study medication.
15. Subjects with inadequate venous access.
16. Subjects vaccinated within 30 days prior to the first dose of study medication. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Subjects will be monitored for 4 days after the one hour infusion. Dose escalation may occur if less than 2 subjects in any cohort of 8 experience DLT.
  Dose limiting toxicity (DLT) will be defined as drug-related grade 2 (moderate) or higher toxicity (excluding fever, chills, nausea or other possible infusion-related effects). The maximum tolerated dose (MTD) will be declared at the dose below which 2 or more subjects experience DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Alam, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Georgoff PE, Nikolian VC, Bonham T, Pai MP, Tafatia C, Halaweish I, To K, Watcharotone K, Parameswaran A, Luo R, Sun D, Alam HB. Safety and Tolerability of Intravenous Valproic Acid in Healthy Subjects: A Phase I Dose-Escalation Trial. Clin Pharmacokinet. 2018 Feb;57(2):209-219. doi: 10.1007/s40262-017-0553-1. PMID 28497259